CLINICAL TRIAL: NCT01606306
Title: Individualized Therapy For Asthma in Toddlers
Acronym: INFANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Principal Investigator, AsthmaNet Data Coordinating Center, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AsthmaNet 004; 1U10HL098115 (NIH)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-01

CONDITIONS: Asthma; Wheezing
Keywords: Asthma; Wheezing; Fluticasone; Montelukast; Preschool-age
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Crossover sequence 1 (Experimental): daily fluticasone propionate, followed by daily montelukast, followed by as needed fluticasone propionate
  Interventions: Drug: daily fluticasone propionate; Drug: Montelukast; Drug: as-needed fluticasone propionate
- Crossover sequence 2 (Experimental): daily fluticasone propionate, followed by as needed fluticasone propionate, followed by daily montelukast
  Interventions: Drug: daily fluticasone propionate; Drug: Montelukast; Drug: as-needed fluticasone propionate
- Crossover sequence 3 (Experimental): daily montelukast, followed by as needed fluticasone propionate, followed by daily fluticasone propionate
  Interventions: Drug: daily fluticasone propionate; Drug: Montelukast; Drug: as-needed fluticasone propionate
- Crossover sequence 4 (Experimental): daily montelukast, followed by daily fluticasone propionate, followed by as needed fluticasone propionate
  Interventions: Drug: daily fluticasone propionate; Drug: Montelukast; Drug: as-needed fluticasone propionate
- Crossover sequence 5 (Experimental): as needed fluticasone propionate, followed by daily fluticasone propionate, followed by daily montelukast
  Interventions: Drug: daily fluticasone propionate; Drug: Montelukast; Drug: as-needed fluticasone propionate
- Crossover sequence 6 (Experimental): as needed fluticasone propionate, followed by daily montelukast, followed by daily fluticasone propionate
  Interventions: Drug: daily fluticasone propionate; Drug: Montelukast; Drug: as-needed fluticasone propionate

INTERVENTIONS:
Drug: daily fluticasone propionate — Flovent® HFA, 44 mcg per inhalation, 2 inhalations twice daily
Drug: Montelukast — Singulair®, 4 mg granules or chewable tablets by mouth once daily in the evening
Drug: as-needed fluticasone propionate — Flovent® HFA, 44 mcg per inhalation, 2 inhalations, as needed for asthma symptoms

SUMMARY:
The INFANT study will test whether, in preschool children 12-59 months of age with persistent asthma, the following Step 2 asthma therapies will provide similar degrees of asthma control:

1. Daily inhaled corticosteroid (ICS) treatment,
2. Daily leukotriene receptor antagonist (LTRA) treatment, and
3. As-needed ICS plus short-acting beta agonist (as-needed ICS/SABA) rescue treatment.

DETAILED DESCRIPTION:
INFANT is a double-blind, randomized clinical trial in which all participants will receive each of the three therapies for 16 weeks by means of a cross-over study design. INFANT aims to determine whether individual children respond better to one treatment than another and, if so, whether those children can be identified by phenotypic characteristics or selected biomarkers. In this regard the INFANT study is expected to address critical gaps in current asthma management guidelines. Ultimately, the findings from this study are expected to help clarify treatment modalities for this population of young preschool children who are extremely difficult to treat.

ELIGIBILITY:
Inclusion Criteria:

* 12-59 months of age.
* If the child is not currently taking long-term asthma controller therapy (meaning that the child has taken no inhaled corticosteroid or leukotriene receptor antagonist medication whatsoever over the past 6 months), then one of the following criteria must be met:

  * Daytime asthma symptoms more than two days per week (average over the past 4 weeks),
  * At least one nighttime awakening from asthma (over the past 4 weeks),
  * Two or more asthma exacerbations requiring systemic corticosteroids in the previous 6 months,
  * Four or more wheezing episodes in the previous 12 months.
* If the child is currently taking long-term asthma controller therapy (meaning that the child has taken daily or intermittent/as-needed inhaled corticosteroid or leukotriene receptor antagonist over the past 6 months), then one of the following criteria must be met:

  * Taking inhaled corticosteroid or leukotriene receptor antagonist for more than 3 months (or more than 90 days) out of the previous 6 months (or 180 days),
  * Daytime asthma symptoms more than two days per week (average over the past 4 weeks),
  * More than one nighttime awakening from asthma (over the past 4 weeks),
  * Two or more asthma exacerbations requiring systemic corticosteroids in the previous 12 months,
  * Four or more wheezing episodes in the previous 12 months.
* Up to date with immunizations, including varicella (unless the subject has already had clinical varicella).
* Willingness to provide informed consent by the child's parent or guardian.

Exclusion Criteria:

* Allergic reaction to the study medications or any component of the study drugs, including (but not limited to) urticaria, rash, angioedema, or hypotension following delivery,
* Chronic medical disorders that could interfere with drug metabolism/excretion (for instance chronic hepatic, biliary, or renal disease),
* Chronic medical disorders that may increase the risk of drug-related injury, including (but not limited to):

  * Osteogenesis imperfecta (increased risk of bone demineralization/fracture with corticosteroid therapy),
  * Crohn's disease, ulcerative colitis, juvenile rheumatoid arthritis, clotting disorders, or Factor deficiency (increased risk of bleeding with corticosteroid therapy),
  * G6PD deficiency (increased risk of hemolytic anemia with acetaminophen use),
  * Phenylketonuria (potential for aspartame exposure with study interventions),
  * Seizure disorder treated with anticonvulsants (risk of acetaminophen toxicity with carbamazepine), or
  * History of clotting disorders or Factor deficiency (increased risk of bleeding with corticosteroids),
* Co-morbid disorders associated with wheezing including (but not limited to) immune deficiency disorders, cystic fibrosis, aspiration, clinically-relevant gastroesophageal reflux, tracheomalacia, congenital airway anomalies (clefts, fistulas, slings, rings), bronchiectasis, bronchopulmonary dysplasia, and/or history of premature birth before 35 weeks gestation,
* Significant developmental delay/failure to thrive, defined as 5th percentile for height and/or weight or crossing of two major percentile lines during the last year for age and sex,
* History of a near-fatal asthma exacerbation requiring intubation or assisted ventilation,
* No primary medical caregiver (e.g., a nurse practitioner, physician assistant, physician, or group medical practice such as a hospital-based clinic) whom the subject can contact for primary medical care,
* Three or more hospitalizations in the previous 12 months for wheezing or respiratory illnesses,
* Treatment with 5 or more courses of systemic corticosteroids (oral, intramuscular or intravenous) in the past 6 months,
* Current use of higher than step 2 NAEPP asthma guideline therapy
* If receiving allergy shots, change in the dose within the past 3 months.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Busse, MD, Study Chair — University of Wisconsin, Madison
Locations (13):
- United States (13):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Children's Hospital & Research Center Oakland, Oakland, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center/Stroger Hospital, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital, Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Rainbow Babies and Children's Hospital, Case Western Reserve University, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Fitzpatrick AM, Jackson DJ, Mauger DT, Boehmer SJ, Phipatanakul W, Sheehan WJ, Moy JN, Paul IM, Bacharier LB, Cabana MD, Covar R, Holguin F, Lemanske RF Jr, Martinez FD, Pongracic JA, Beigelman A, Baxi SN, Benson M, Blake K, Chmiel JF, Daines CL, Daines MO, Gaffin JM, Gentile DA, Gower WA, Israel E, Kumar HV, Lang JE, Lazarus SC, Lima JJ, Ly N, Marbin J, Morgan W, Myers RE, Olin JT, Peters SP, Raissy HH, Robison RG, Ross K, Sorkness CA, Thyne SM, Szefler SJ; NIH/NHLBI AsthmaNet. Individualized therapy for persistent asthma in young children. J Allergy Clin Immunol. 2016 Dec;138(6):1608-1618.e12. doi: 10.1016/j.jaci.2016.09.028. Epub 2016 Oct 21. PMID 27777180

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3 | Crossover Sequence 4 | Crossover Sequence 5 | Crossover Sequence 6
Started | 50 | 49 | 51 | 51 | 52 | 47
Completed First Treatment Period | 43 | 47 | 47 | 45 | 47 | 44
Completed Second Treatment Period | 41 | 38 | 43 | 44 | 46 | 41
Completed Third Treatment Period | 35 | 39 | 37 | 38 | 41 | 36
Completed | 35 | 39 | 37 | 38 | 41 | 36
Not Completed | 15 | 10 | 14 | 13 | 11 | 11
Not completed — Lack of Efficacy | 2 | 1 | 4 | 4 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 2 | 0
Not completed — Lost to Follow-up | 7 | 4 | 5 | 4 | 3 | 5
Not completed — Withdrawal by Subject | 4 | 3 | 4 | 4 | 5 | 4
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3 | Crossover Sequence 4 | Crossover Sequence 5 | Crossover Sequence 6 | Total
Number analyzed (Participants) | 50 | 49 | 51 | 51 | 52 | 47 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 49 | 51 | 51 | 52 | 47 | 300
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 38.3 (13.6) | 40.7 (12.4) | 38.7 (11.6) | 38.6 (15.1) | 41.7 (12.7) | 41.2 (14.0) | 39.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 19 | 21 | 18 | 23 | 121
  Male | 30 | 29 | 32 | 30 | 34 | 24 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 12 | 10 | 11 | 12 | 10 | 72
  Not Hispanic or Latino | 33 | 37 | 41 | 40 | 40 | 37 | 228
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2 | 0 | 1 | 5
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Black or African American | 11 | 15 | 20 | 13 | 20 | 18 | 97
  White | 25 | 27 | 24 | 30 | 21 | 21 | 148
  More than one race | 10 | 6 | 7 | 5 | 10 | 7 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 49 | 51 | 51 | 52 | 47 | 300
Parental Asthma [Number; unit: participants]
  Present | 30 | 29 | 29 | 32 | 35 | 23 | 178
  Not Present | 20 | 20 | 22 | 19 | 17 | 24 | 122
Systemic corticosteroids in past 12 monts [Number; unit: participants]
  Used | 37 | 35 | 37 | 40 | 39 | 36 | 224
  Not used | 13 | 14 | 14 | 11 | 13 | 11 | 76
Hospitalized in past 12 months [Number; unit: participants]
  Hospitalized | 9 | 14 | 11 | 6 | 13 | 12 | 65
  Not hospitalized | 41 | 35 | 40 | 45 | 39 | 35 | 235
Allergen Test [Number; unit: participants]
  Positive test | 18 | 20 | 20 | 21 | 25 | 17 | 121
  Negative test | 32 | 29 | 31 | 30 | 27 | 30 | 179
Eczema [Number; unit: participants]
  Present | 21 | 28 | 27 | 28 | 26 | 30 | 160
  Not Present | 29 | 21 | 24 | 23 | 26 | 17 | 140
Blood eosinophils [Median (Inter-Quartile Range); unit: number of cells per micro-liter] | 183 [111 to 435] | 234 [153 to 572] | 258 [133 to 460] | 255 [175 to 457] | 308 [184 to 496] | 310 [182 to 536] | 258 [158 to 492]
Serum IgE [Median (Inter-Quartile Range); unit: international units per liter] | 67 [25 to 212] | 106.5 [22 to 463] | 64 [21 to 141] | 64 [31 to 143] | 87 [19 to 237] | 84 [19 to 348] | 70 [22 to 208]

OUTCOME MEASURES:

1. Primary Outcome: Differential Response to the Three Therapies Based on Fixed Threshold Criteria for the Following Asthma Control Measures: Use of Oral Prednisone for Acute Asthma Exacerbations and Asthma Control Days.
Description: The primary outcome was differential response to the three therapies on the basis of fixed threshold criteria for the following asthma control measures, which encompassed domains of risk and impairment: the time from the start of the treatment period to an asthma exacerbation treated with systemic corticosteroids, and the annualized number of asthma control days (ACDs) from within that period. ACDs were defined as full calendar days without symptoms, rescue medication use, or unscheduled healthcare visits. Children were defined as differential responders if, first, the time to an asthma exacerbation was at least four weeks longer, or second, if the number of annualized ACDs was at least 31 days more for one treatment than another, in that order. If neither threshold was met, the participant was considered a non differential responder. Differential response was determined in children completing at least two treatment periods and at least 50% of the daily diary entries for each period.
Time Frame: The last 14 weeks of each 16-week treatment period
Population: Differential response was determined in children completing at least two treatment periods and at least 50% of the daily diary entries for each period.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- All Evaluable Participants: Differential response was determined in children completing at least two treatment periods and at least 50% of the daily diary entries for each period. Because placebo washouts were not performed, the data collected during the first two weeks of each period were not included in the analysis of ACDs. Days with missing diary data were also excluded from ACD determination.
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 230
probability
  Non-differential responders | .26 [.26 to .26]
  Responded best to daily ICS | .40 [.33 to .47]
  Responded best to daily LTRA | .18 [.13 to .23]
  Responded best to as-needed ICS | .16 [.11 to .21]
Statistical Analysis 1: Comparison: All Evaluable Participants; The primary analysis tested the null hypothesis of all three treatments having equal probability to yield the best response as defined by the criteria defining the primary outcome. A sample size of 300 participants was selected to test the primary null hypothesis of all three treatments having equal probability (one-third) to yield the best response with statistical power of at least 0.90 if any one of the three treatments actually has probability of at least one-half to yield the best response; Test type: Superiority or Other; p < 0.0001, rank-order logistic regression — Rank-ordered logistic regression (ROLR) was used to model the probability of best response for each treatment and bootstrapping was used to calculate confidence intervals; ROLR is in the class of Discrete Choice models, which seek to estimate the probability that an individual responds best to a specific treatments; The probabilistic construct of the Discrete Choice (DC) model does not reflect individual behavior that is intrinsically probabilistic, but rather population heterogeneity. DC models rely on stochastic assumptions to account for unobserved factors related to the treatments themselves and to characteristics of study participants. Specifically, that each treatment has an underlying utility that may differ from one individual to another. Mathematically, these utilities are represented by U_t, where t denotes the treatment. Utility can be thought of as a latent variable quantifying treatment response where higher values indicate better response. The U_t can be used to find the probability (P) of best response for each treatment by the following equation: P_t = exp(U_t) / [exp(U_A) + exp(U_B) + exp(U_C)], where A, B, and C, denote the three study treatments. The primary analysis tested whether the three treatments have equal utility and, thus, equal probability of best response

ADVERSE EVENTS:
Groups:
- Daily ICS: Daily inhaled corticosteroid (ICS) treatment
- As-needed ICS: As-needed ICS plus short-acting beta agonist (as-needed ICS/SABA) rescue treatment.
- Daily LTRA: Daily leukotriene receptor antagonist (LTRA) treatment
Arm/Group | Daily ICS | As-needed ICS | Daily LTRA
Serious Adverse Events (participants affected / at risk) | 2/300 | 8/300 | 8/300
Other Adverse Events (participants affected / at risk) | 212/300 | 206/300 | 212/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily ICS (N=300) | As-needed ICS (N=300) | Daily LTRA (N=300)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Simple laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Penumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 8 (8)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
tonsilitis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily ICS (N=300) | As-needed ICS (N=300) | Daily LTRA (N=300)
Otitis media (Ear and labyrinth disorders) | 22 (27) | 24 (27) | 28 (29)
Fever (General disorders) | 100 (127) | 89 (111) | 109 (146)
Headache (General disorders) | 16 (20) | 14 (17) | 11 (17)
Acute upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 39 (45) | 41 (53) | 54 (65)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 16 (21) | 26 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (31) | 35 (42) | 26 (32)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 41 (47) | 59 (70) | 68 (84)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No